CLINICAL TRIAL: NCT02583048
Title: A Trial of the Safety, Tolerability, and Pharmacokinetics of Bedaquiline and Delamanid, Alone and in Combination, Among Participants Taking Multidrug Treatment for Drug-Resistant Pulmonary Tuberculosis
Brief Title: Evaluating the Safety, Tolerability, and Pharmacokinetics of Bedaquiline and Delamanid, Alone and in Combination, For Drug-Resistant Pulmonary Tuberculosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5343; 12005 (Registry Identifier: DAIDS-ES Registry)
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Results first posted 2020-01-29 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Tuberculosis; HIV Infections
MeSH Terms: conditions — Tuberculosis; HIV Infections | interventions — bedaquiline; OPC-67683; dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1: Bedaquiline (Experimental): Participants received 400 mg of bedaquiline once a day for 2 weeks followed by 200 mg of bedaquiline three times a week for 22 weeks.
  Participants also received Multidrug Background Treatment (MBT) for TB.
  For HIV-positive participants only, one 50 mg tablet of Dolutegravir was taken in combination with two NRTIs until study completion.
  Interventions: Drug: Bedaquiline; Drug: Dolutegravir; Drug: Multidrug Background Treatment (MBT) for TB
- Arm 2: Delamanid (Experimental): Participants received 100 mg of delamanid twice a day for 24 weeks.
  Participants also received Multidrug Background Treatment (MBT) for TB.
  For HIV-positive participants only, one 50 mg tablet of Dolutegravir was taken in combination with two NRTIs until study completion.
  Interventions: Drug: Delamanid; Drug: Dolutegravir; Drug: Multidrug Background Treatment (MBT) for TB
- Arm 3: Bedaquiline and Delamanid (Experimental): Participants received 400 mg of bedaquiline once a day and 100 mg of delamanid twice a day for 2 weeks. They then received 200 mg of bedaquiline three times a week and 100 mg of delamanid twice a day for 22 weeks.
  Participants also received Multidrug Background Treatment (MBT) for TB.
  For HIV-positive participants only, one 50 mg tablet of Dolutegravir was taken in combination with two NRTIs until study completion.
  Interventions: Drug: Bedaquiline; Drug: Delamanid; Drug: Dolutegravir; Drug: Multidrug Background Treatment (MBT) for TB

INTERVENTIONS:
Drug: Bedaquiline — Four 100 mg tablets (400 mg) orally once a day for 2 weeks, followed by two 100 mg tablets (200 mg) orally three times a week for 22 weeks.
  Other Names: Sirturo
  Arms: Arm 1: Bedaquiline; Arm 3: Bedaquiline and Delamanid
Drug: Delamanid — Two 50 mg tablets (100 mg) orally with food twice a day for 24 weeks.
  Other Names: Deltyba
  Arms: Arm 2: Delamanid; Arm 3: Bedaquiline and Delamanid
Drug: Dolutegravir — For HIV-positive participants only: one 50 mg tablet orally once daily, to be used in combination with two NRTIs until study completion. (NRTIs were not provided by the study.)
  Other Names: Tivicay
Drug: Multidrug Background Treatment (MBT) for TB — A standardized MBT regimen for MDR- or RR-TB except in cases where a participant had known resistance to one of the components of local standard treatment. MBT was provided by the local program.

SUMMARY:
This study evaluated the safety, tolerability, and pharmacokinetics of the anti-tuberculosis (TB) drugs bedaquiline (BDQ) and delamanid (DLM), alone and in combination, among participants (with or without HIV co-infection) taking multidrug treatment for multidrug-resistant tuberculosis (MDR-TB) or rifampin-monoresistant TB (RR-TB).

DETAILED DESCRIPTION:
Bedaquiline (BDQ) and delamanid (DLM) are two newly approved anti-TB drugs and are both well tolerated. However, the combined effect of these two drugs has not been studied. Combining these two drugs, together with other anti-TB drugs, may improve outcomes for people with MDR-TB or RR-TB. The purpose of this study was to evaluate the safety, tolerability, and pharmacokinetics of BDQ and DLM, alone and in combination, among participants (with or without HIV co-infection) taking multidrug treatment for MDR-TB or RR-TB, and specifically to evaluate the effect of these drugs on the heart.

Participants were randomly assigned to one of three arms: participants in Arm 1 received BDQ, participants in Arm 2 received DLM, and participants in Arm 3 received BDQ and DLM. All participants received their assigned study drugs for 24 weeks together with multidrug background treatment (MBT) for MDR-TB or RR-TB (not provided by the study). HIV-infected participants also received dolutegravir, to be used in combination with two nucleoside reverse transcriptase inhibitors (NRTIs) until study completion. NRTIs were not provided by the study. At study entry participants were initially required to be hospitalized for 2 months, however after an interim analysis, the period of hospitalization was shortened to 2 weeks.

Study visits occurred at entry, each week for 8 weeks after study entry, every other week until week 24, and at weeks 28, 36, 48, 60, 72, 84, 96 and 128. Visits included physical examinations, blood collection, urine collection, sputum sample collection, hair sample collection, chest x-rays, pregnancy testing, electrocardiograms (ECGs), and adherence questionnaires.

Participants were also asked to take part in an optional cerebrospinal fluid sampling study that entailed a lumbar puncture, to be done at weeks 8 or 24.

ELIGIBILITY:
Inclusion Criteria:

* Documented pulmonary infection due to strains of MTB with (a) resistance to isoniazid (INH) and rifampin (RIF) (MDR-TB) or (b) resistance to RIF but not INH (RR-TB) from a sputum sample collected within 60 days prior to entry.
* Laboratory confirmation of infection with an MTB strain that is susceptible to fluoroquinolones and aminoglycosides within 60 days prior to entry.
* HIV-1 infection status documented as either absent or present, as defined below:

  * Absence of HIV-1 infection, within 60 days prior to entry. OR
  * HIV-1 infection
* For HIV-positive participants only: CD4+ count greater than or equal to 100 cells/mm^3 within 60 days prior to entry.
* For HIV-positive participants only: For participants on ART for greater than or equal to 6 months and have an HIV-1 viral load greater than 500 copies/mL within 60 days prior to entry, a HIV-1 genotype within 60 days prior to entry must have shown that at least one fully active NRTI was available to the participant within the country program.
* For females of reproductive potential, a negative serum pregnancy test within 48 hours prior to entry
* All participants of reproductive potential who are participating in sexual activity that could lead to pregnancy must have agreed to use one method of birth control while receiving TB study medications and for 6 months after stopping TB study medications.
* Participants who were not of reproductive potential were eligible without requiring the use of contraceptives.
* For HIV-positive female participants of reproductive potential, the use of contraceptives was required for the full duration of time the participant was taking dolutegravir (ie, through study completion at week 128).
* Chest x-ray performed within 60 days prior to entry to classify participant as having cavitary or non-cavitary disease
* Documentation of Karnofsky performance score greater than or equal to 50 within 14 days prior to study entry
* Ability and willingness of participant or legally authorized representative to provide informed consent
* Willingness to be hospitalized for the required inpatient component of the study
* Taking MBT for a minimum of 7 days within the 10 days prior to entry

Exclusion Criteria:

* History of clinically relevant, currently active or underlying gastrointestinal, hepatic, cardiovascular, nervous system, psychiatric, metabolic (e.g., untreated hypothyroidism), renal, respiratory (other than due to TB), inflammatory, neoplastic, skin, immunological or infectious disease, which is not stable and controlled, that in the opinion of the investigator would preclude safe participation in the trial
* Current clinically relevant extrapulmonary TB, in the opinion of the site investigator, including but not limited to central nervous system (CNS) TB or TB osteoarthritis
* Previous treatment for MDR- or RR-TB, other than for the qualifying episode, at any time in the past
* Receipt of BDQ or DLM at any time in the past
* Breastfeeding
* QTcF interval greater than 450 ms within 72 hours prior to entry
* Clinically significant ECG abnormality in the opinion of the site investigator within 60 days prior to entry, including but not limited to second or third degree atrioventricular (AV) block, prolongation of the QRS complex over 120 ms (in both male and female participants), or clinically important arrhythmia
* Current clinically relevant cardiovascular disorder in the opinion of the site investigator, including but not limited to heart failure, coronary heart disease, arrhythmia, or tachyarrhythmia
* Known family history of Long QT Syndrome in a first-degree relative (i.e., parent, offspring, or sibling)
* Requirement or expected requirement for protease inhibitors (PIs), efavirenz (EFV), or any other medication that is a moderate to strong inhibitor or inducer of CYP3A and CYP3A4 over the 24 weeks of study treatment. NOTE: Participants taking a PI or EFV can be switched to a treatment that is allowed in the study, but the PI must be stopped at least 2 days prior to starting study MDR- or RR-TB drugs and EFV must be stopped at least 7 days prior to starting study MDR- or RR-TB drugs.
* Requirement or expected requirement for a medication that significantly prolongs QTc, including but not limited to moxifloxacin (levofloxacin is acceptable), from 72 hours prior to study entry through 4 weeks after discontinuation of study treatment (week 28)
* Requirement or expected requirement of clofazimine, from 7 days prior to study entry through week 24 (discontinuation of study treatment).
* For individuals receiving the WHO short course regimen that contains clofazimine, receipt of more than 21 cumulative days of clofazimine at any time prior to, or at the time of, study entry.
* Known allergy/sensitivity or any hypersensitivity to components of study TB drugs or their formulation or to the nitroimidazole class of antibiotics
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Any of the following laboratory abnormalities within 14 days prior to entry:

  1. Serum creatinine greater than 1.4 x upper limit of normal (ULN)
  2. Lipase greater than 1.6 x ULN
  3. Alanine aminotransferase (ALT) greater than 2.5 x ULN
  4. Total bilirubin greater than 1.6 x ULN
  5. Potassium less than 3.4 or greater than 5.6 mmol/L; magnesium less than 0.59 mmol/L; calcium less than 1.75 mmol/L
* Known current hepatitis B or C infection, current treatment for hepatitis B or hepatitis C infection, or positive for hepatitis B surface antigen or hepatitis C antibodies within 60 days prior to entry
* Among participants with HIV infection, in whom use of dolutegravir (DTG) is anticipated, any of the following:

  1. Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, esophageal varices, or persistent jaundice), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
  2. History or presence of allergy to DTG or its components
  3. Severe hepatic impairment (Class C) as determined by Child-Pugh classification
  4. Previous use of raltegravir
* Documentation of any new and/or unstable AIDS-defining illness (other than TB) as defined by the CDC within 60 days prior to entry
* Acute or serious illness (other than TB) requiring systemic treatment and/or hospitalization within 60 days prior to entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2021-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Dooley, MD, PhD, Study Chair — Johns Hopkins Adult AIDS CRS; Gary Maartens, MBChB, MMed, Study Chair — University of Cape Town
Locations (3):
- Barranco CRS, Lima, Peru
- South Africa (2):
  - Task Applied Science (TASK) CRS, Cape Town, Western Cape
  - South African Tuberculosis Vaccine Initiative (SATVI) CRS, Cape Town, Western Cape

REFERENCES:
- [Derived] Tanneau L, Karlsson MO, Diacon AH, Shenje J, De Los Rios J, Wiesner L, Upton CM, Dooley KE, Maartens G, Svensson EM. Population Pharmacokinetics of Delamanid and its Main Metabolite DM-6705 in Drug-Resistant Tuberculosis Patients Receiving Delamanid Alone or Coadministered with Bedaquiline. Clin Pharmacokinet. 2022 Aug;61(8):1177-1185. doi: 10.1007/s40262-022-01133-2. Epub 2022 Jun 7. PMID 35668346
- [Derived] Dooley KE, Rosenkranz SL, Conradie F, Moran L, Hafner R, von Groote-Bidlingmaier F, Lama JR, Shenje J, De Los Rios J, Comins K, Morganroth J, Diacon AH, Cramer YS, Donahue K, Maartens G; AIDS Clinical Trials Group (ACTG) A5343 DELIBERATE Study Team. QT effects of bedaquiline, delamanid, or both in patients with rifampicin-resistant tuberculosis: a phase 2, open-label, randomised, controlled trial. Lancet Infect Dis. 2021 Jul;21(7):975-983. doi: 10.1016/S1473-3099(20)30770-2. Epub 2021 Feb 12. PMID 33587897
- See also: Location of DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.0, November 2014 — http://rsc.tech-res.com/clinical-research-sites/safety-reporting/daids-grading-tables
- See also: Location of Version 2.0 the DAIDS EAE Manual for Expedited AE Reporting — http://rsc.tech-res.com/clinical-research-sites/safety-reporting/manual

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from August 2016 to July 2018 at 3 non-US clinical research sites.
Pre-assignment Details: Participants were randomized with equal probability to each of the 3 experimental arms.
Groups:
- Arm 1: Bedaquiline: Participants received 400 mg of bedaquiline once a day for 2 weeks followed by 200 mg of bedaquiline three times a week for 22 weeks.
  For HIV-positive participants only: One 50 mg tablet of Dolutegravir was taken orally once daily, to be used in combination with two NRTIs until study completion. (NRTIs not provided by the study.)
  Participants also took Multidrug Background Treatment (MBT) for TB (not provided by the study).
- Arm 2: Delamanid: Participants received 100 mg of delamanid twice a day for 24 weeks.
  For HIV-positive participants only: One 50 mg tablet of Dolutegravir was taken orally once daily, to be used in combination with two NRTIs until study completion. (NRTIs not provided by the study.)
  Participants also took Multidrug Background Treatment (MBT) for TB (not provided by the study).
- Arm 3: Bedaquiline and Delamanid: Participants received 400 mg of bedaquiline once a day and 100 mg of delamanid twice a day for 2 weeks. They then received 200 mg of bedaquiline three times a week and 100 mg of delamanid twice a day for 22 weeks.
  For HIV-positive participants only: One 50 mg tablet of Dolutegravir was taken orally once daily, to be used in combination with two NRTIs until study completion. (NRTIs not provided by the study.)
  Participants also took Multidrug Background Treatment (MBT) for TB (not provided by the study).
Period: Overall Study
Arm/Group | Arm 1: Bedaquiline | Arm 2: Delamanid | Arm 3: Bedaquiline and Delamanid
Started | 28 | 28 | 28
Completed | 28 | 27 | 27
Not Completed | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Failed to meet eligibility criterion | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Bedaquiline | Arm 2: Delamanid | Arm 3: Bedaquiline and Delamanid | Total
Number analyzed (Participants) | 28 | 28 | 28 | 84
Age, Continuous [Median (Full Range); unit: years] | 34.5 [20 to 58] | 32 [18 to 73] | 34 [18 to 55] | 34 [18 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 8 | 21
  Male | 22 | 21 | 20 | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 0 | 1 | 0 | 1
  Black African | 16 | 11 | 11 | 38
  Mestizo | 1 | 2 | 3 | 6
  Coloured | 11 | 13 | 14 | 38
  Other | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 27 | 26 | 25 | 78
  Peru | 1 | 2 | 3 | 6
Baseline QTcF [Median (Full Range); unit: milliseconds] | 394.3 [360.7 to 461.0] | 406.2 [364.3 to 445.0] | 387.3 [368.3 to 422.3] | 395.5 [360.7 to 461.0]
HIV-1 Positive [Count of Participants; unit: Participants] | 10 | 11 | 10 | 31

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in QTcF
Description: Mean change from baseline in QTcF (ie, QTcF prolongation) in milliseconds (ms), where baseline QTcF was represented by QTcF durations measured at week 0, and post-baseline QTcF was represented by QTcF durations measured at weeks 8 through 24 (pooled). QTcF calculated as average of 1-3 available QTcF values per visit.
Time Frame: Baseline and at weeks 8, 10, 12, 14, 16, 18, 20, 22 and 24
Population: Participants with a baseline QTcF measurement, and at least one post-baseline QTcF measurement from a visit conducted at week 8 through 24, prior to permanent discontinuation of study Tuberculosis (TB) drug and without a temporary discontinuation of study TB drug of 7 or more days immediately preceding the measurement.
Measure: Mean (95.1% Confidence Interval); unit: milliseconds (ms)
Groups:
- Arm 1: Bedaquiline: Participants received 400 mg of bedaquiline once a day for 2 weeks followed by 200 mg of bedaquiline three times a week for 22 weeks.
  For HIV-positive participants only: dolutegravir was administered at a dose of one 50 mg tablet once daily, to be used in combination with two NRTIs until study completion. (NRTIs not provided by the study.)
  Participants also took Multidrug Background Treatment (MBT) for TB (not provided by the study).
- Arm 2: Delamanid: Participants received 100 mg of delamanid twice a day for 24 weeks.
  For HIV-positive participants only: dolutegravir was administered at a dose of one 50 mg tablet once daily, to be used in combination with two NRTIs until study completion. (NRTIs not provided by the study.)
  Participants also took Multidrug Background Treatment (MBT) for TB (not provided by the study).
- Arm 3: Bedaquiline and Delamanid: Participants received 400 mg of bedaquiline once a day and 100 mg of delamanid twice a day for 2 weeks. They then received 200 mg of bedaquiline three times a week and 100 mg of delamanid twice a day for 22 weeks.
  For HIV-positive participants only: dolutegravir was administered at a dose of one 50 mg tablet once daily, to be used in combination with two NRTIs until study completion. (NRTIs not provided by the study.)
  Participants also took Multidrug Background Treatment (MBT) for TB (not provided by the study).
Arm/Group | Arm 1: Bedaquiline | Arm 2: Delamanid | Arm 3: Bedaquiline and Delamanid
Number analyzed (Participants) | 26 | 25 | 24
milliseconds (ms) | 12.3 [7.8 to 16.7] | 8.6 [4.0 to 13.1] | 20.7 [16.1 to 25.3]
Statistical Analysis 1: Comparison: Arm 1: Bedaquiline vs Arm 3: Bedaquiline and Delamanid; Test type: Superiority; Mean Difference (Net) = 8.4, 95.1% CI 2-sided [2.0 to 14.8] — Arm 3 minus Arm 1 difference in change from baseline estimated from ANOVA model. Interim analysis conducted when week 24 QT data was available for ≥12 participants stipulated 99.9% confidence interval; original coverage of 95% was widened to 95.1%
Statistical Analysis 2: Comparison: Arm 2: Delamanid vs Arm 3: Bedaquiline and Delamanid; Test type: Superiority; Mean Difference (Net) = 12.1, 95.1% CI 2-sided [5.7 to 18.6] — Arm 3 minus Arm 2 difference in change from baseline estimated from ANOVA model. Interim analysis conducted when week 24 QT data was available for ≥12 participants stipulated 99.9% confidence interval; original coverage of 95% was widened to 95.1%

2. Primary Outcome: Post-Baseline QTcF
Description: Baseline and post-baseline absolute QTcF in milliseconds (ms) estimated using an ANOVA model, where baseline QTcF was represented by QTcF durations measured at week 0, and post-baseline QTcF was represented by QTcF durations measured at weeks 8 through 24 (pooled). QTcF calculated as average of 1-3 available QTcF values per visit. Interim analysis conducted when week 24 QT data was available for ≥12 participants stipulated 99.9% confidence interval; original coverage of 95% was widened to 95.1%.
Time Frame: Baseline and at weeks 8, 10, 12, 14, 16, 18, 20, 22, and 24.
Population: as for outcome 1
Measure: Least Squares Mean (95.1% Confidence Interval); unit: milliseconds (ms)
Arm/Group | Arm 1: Bedaquiline | Arm 2: Delamanid | Arm 3: Bedaquiline and Delamanid
Number analyzed (Participants) | 26 | 25 | 24
milliseconds (ms)
  Baseline | 397.4 [389.3 to 405.6] | 404.9 [396.6 to 413.2] | 391.7 [383.2 to 400.2]
  Post-baseline | 409.7 [402.5 to 416.8] | 413.4 [406.1 to 420.8] | 412.4 [405.0 to 419.9]

3. Secondary Outcome: Percentage of Participants With an Occurrence of QTcF Greater Than 500 Milliseconds (ms)
Description: Participants who experienced QTcF greater than 500 ms at least once at any time from week 2 to 24. QTcF calculated as average of 1-3 available QTcF values per visit.
Time Frame: At weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22 and 24
Population: Participants who took at least one dose of study TB treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: Bedaquiline | Arm 2: Delamanid | Arm 3: Bedaquiline and Delamanid
Number analyzed (Participants) | 28 | 27 | 27
Percentage of participants | 0 [0 to 12] | 0 [0 to 13] | 0 [0 to 13]

4. Secondary Outcome: Percentage of Participants With an Increase in QTcF From Baseline of Greater Than 60 Milliseconds (ms)
Description: Participants who experienced QTcF increase from baseline greater than 60 ms at least once at any time from week 2 to 24. QTcF calculated as average of 1-3 available QTcF values per visit.
Time Frame: Baseline and at weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22 and 24
Population: Participants who took at least one dose of study TB treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: Bedaquiline | Arm 2: Delamanid | Arm 3: Bedaquiline and Delamanid
Number analyzed (Participants) | 28 | 27 | 27
Percentage of participants | 4 [0 to 18] | 0 [0 to 13] | 7 [1 to 24]

5. Secondary Outcome: Changes in QTcF From Baseline
Description: Change from baseline in QTcF, calculated as the difference between each post-baseline week and week 0. (QTcF calculated as average of 1-3 available QTcF values per visit.)
Time Frame: Baseline and at weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 and 28.
Population: Participants with baseline and at least one post baseline QTcF collected at a scheduled visit while taking study TB drug(s).
Measure: Median (Full Range); unit: milliseconds (ms)
Arm/Group | Arm 1: Bedaquiline | Arm 2: Delamanid | Arm 3: Bedaquiline and Delamanid
Number analyzed (Participants) | 28 | 26 | 26
milliseconds (ms)
  Change from baseline to Week 2: number analyzed (Participants) | 27 | 26 | 26
  Change from baseline to Week 2 | 16.70 [-25.70 to 57.00] | 4.15 [-25.70 to 24.30] | 13.15 [-6.70 to 55.70]
  Change from baseline to Week 4: number analyzed (Participants) | 28 | 25 | 25
  Change from baseline to Week 4 | 15.00 [-21.00 to 40.70] | 8.70 [-15.70 to 24.70] | 14.30 [-8.70 to 50.30]
  Change from baseline to Week 6: number analyzed (Participants) | 26 | 25 | 25
  Change from baseline to Week 6 | 15.30 [-25.30 to 40.00] | 9.30 [-19.00 to 37.70] | 15.30 [-11.00 to 33.70]
  Change from baseline to Week 8: number analyzed (Participants) | 26 | 25 | 25
  Change from baseline to Week 8 | 12.00 [-40.30 to 47.30] | 7.00 [-30.30 to 39.00] | 20.30 [-14.00 to 47.30]
  Change from baseline to Week 10: number analyzed (Participants) | 25 | 24 | 23
  Change from baseline to Week 10 | 10.30 [-30.30 to 51.00] | 7.80 [-25.30 to 37.70] | 18.30 [-15.00 to 58.30]
  Change from baseline to Week 12: number analyzed (Participants) | 25 | 23 | 25
  Change from baseline to Week 12 | 9.30 [-11.70 to 46.30] | 10.30 [-21.00 to 38.70] | 20.30 [-20.30 to 50.30]
  Change from baseline to Week 14: number analyzed (Participants) | 25 | 23 | 25
  Change from baseline to Week 14 | 12.70 [-16.00 to 53.00] | 5.30 [-18.00 to 49.00] | 21.30 [-19.00 to 51.00]
  Change from baseline to Week 16: number analyzed (Participants) | 24 | 20 | 24
  Change from baseline to Week 16 | 15.35 [-34.30 to 55.30] | 7.35 [-46.00 to 38.70] | 21.00 [-22.70 to 62.70]
  Change from baseline to Week 18: number analyzed (Participants) | 24 | 21 | 23
  Change from baseline to Week 18 | 17.65 [-17.30 to 72.30] | 11.70 [-28.30 to 39.30] | 12.70 [-26.70 to 66.30]
  Change from baseline to Week 20: number analyzed (Participants) | 25 | 22 | 24
  Change from baseline to Week 20 | 9.30 [-24.30 to 46.70] | 13.65 [-21.30 to 29.30] | 21.00 [-18.30 to 70.00]
  Change from baseline to Week 22: number analyzed (Participants) | 24 | 22 | 24
  Change from baseline to Week 22 | 12.00 [-16.00 to 56.70] | 9.00 [-15.70 to 34.30] | 20.85 [-19.30 to 75.00]
  Change from baseline to Week 24: number analyzed (Participants) | 25 | 22 | 23
  Change from baseline to Week 24 | 11.70 [-26.00 to 46.00] | 13.00 [-19.30 to 40.30] | 24.00 [-19.00 to 46.30]
  Change from baseline to Week 28: number analyzed (Participants) | 25 | 19 | 22
  Change from baseline to Week 28 | 13.30 [-20.30 to 43.00] | 6.00 [-25.30 to 38.30] | 17.65 [-16.00 to 55.70]

6. Secondary Outcome: Percentage of Participants With an Occurrence of QTcF >480 and ≤500 Milliseconds (ms)
Description: Participants who experienced QTcF >480 and ≤500 ms at least once at any time from week 2 to 24. QTcF calculated as average of 1-3 available QTcF values per visit.
Time Frame: At weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22 and 24
Population: Participants who took at least one dose of study TB drug(s).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: Bedaquiline | Arm 2: Delamanid | Arm 3: Bedaquiline and Delamanid
Number analyzed (Participants) | 28 | 27 | 27
Percentage of participants | 0 [0 to 12] | 0 [0 to 13] | 0 [0 to 13]

7. Secondary Outcome: Percentage of Participants With an Occurrence of QTcF Increase From Baseline of >30 and ≤60 Milliseconds (ms)
Description: Participants who experienced QTcF increase from baseline of >30 and ≤60 ms at least once at any time from week 2 to 24. QTcF calculated as average of 1-3 available QTcF values per visit.
Time Frame: Baseline and at weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22 and 24
Population: Participants who took at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: Bedaquiline | Arm 2: Delamanid | Arm 3: Bedaquiline and Delamanid
Number analyzed (Participants) | 28 | 27 | 27
Percentage of participants | 32 [16 to 52] | 41 [22 to 61] | 37 [19 to 58]

8. Secondary Outcome: BDQ PK Parameter Minimum Plasma Concentration (Cmin) Determined Based on BDQ Levels From Individual Participants Enrolled in Arms 1 and 3
Description: This evaluates the effect of DLM on the BDQ PK parameter Cmin obtained from participants enrolled in Arms 1 and 3 (without and with co-administration of DLM). Cmin defines minimum concentration observed over the first 22 hours of the BDQ dosing interval.
Time Frame: Intensive BDQ PK samples at pre-dose, 5h, 7h, 10h and 22h post-dose at weeks 2, 8 and 24
Population: Participants who took at least one dose of study treatment, and were taking study drug at the time of the PK visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1: Bedaquiline | Arm 3: Bedaquiline and Delamanid
Number analyzed (Participants) | 28 | 24
ng/mL
  Week 2 | 796.8 (406.1) | 850.9 (343.8)
  Week 8: number analyzed (Participants) | 25 | 21
  Week 8 | 505.9 (218.6) | 601.9 (212.6)
  Week 24: number analyzed (Participants) | 24 | 18
  Week 24 | 653.4 (271.3) | 629.4 (247.0)
Statistical Analysis 1: Comparison: Arm 1: Bedaquiline vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 2; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 1.117, 90% CI 2-sided [0.884 to 1.411] — The numerator represents Arm 3 and the denominator represents Arm 1
Statistical Analysis 2: Comparison: Arm 1: Bedaquiline vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 8; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 1.202, 90% CI 2-sided [0.989 to 1.461] — The numerator represents Arm 3 and the denominator represents Arm 1
Statistical Analysis 3: Comparison: Arm 1: Bedaquiline vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 24; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 0.958, 90% CI 2-sided [0.774 to 1.187] — The numerator represents Arm 3 and the denominator represents Arm 1

9. Secondary Outcome: BDQ PK Parameter Maxmum Plasma Concentration (Cmax) Determined Based on BDQ Levels From Individual Participants Enrolled in Arms 1 and 3
Description: This evaluates the effect of DLM on the BDQ PK parameter Cmax obtained from participants enrolled in Arms 1 and 3 (without and with co-administration of DLM). Cmax defines maximum concentration observed over the first 22 hours of the BDQ dosing interval.
Time Frame: Intensive BDQ PK samples at pre-dose, 5h, 7h, 10h and 22h post-dose at weeks 2, 8 and 24
Population: Participants who took at least one dose of study treatment, and were taking study drug at the time of the PK visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1: Bedaquiline | Arm 3: Bedaquiline and Delamanid
Number analyzed (Participants) | 28 | 24
ng/mL
  Week 2 | 2434.3 (1148.4) | 2405.2 (1128.2)
  Week 8: number analyzed (Participants) | 25 | 21
  Week 8 | 1455.6 (670.6) | 1477.2 (704.7)
  Week 24: number analyzed (Participants) | 24 | 18
  Week 24 | 1507.3 (495.8) | 1368.2 (518.6)
Statistical Analysis 1: Comparison: Arm 1: Bedaquiline vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 2; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 0.986, 90% CI 2-sided [0.801 to 1.215] — The numerator represents Arm 3 and the denominator represents Arm 1
Statistical Analysis 2: Comparison: Arm 1: Bedaquiline vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 8; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 0.978, 90% CI 2-sided [0.764 to 1.251] — The numerator represents Arm 3 and the denominator represents Arm 1
Statistical Analysis 3: Comparison: Arm 1: Bedaquiline vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 24; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 0.859, 90% CI 2-sided [0.667 to 1.108] — The numerator represents Arm 3 and the denominator represents Arm 1

10. Secondary Outcome: BDQ PK Parameter Area Under the Concentration Time Curve (AUC 0-22h) Calculated Based on Intensive PK Samples Obtained From Individual Participants Enrolled in Arms 1 and 3
Description: This evaluates the effect of DLM on the BDQ PK parameter AUC 0-22h obtained from participants enrolled in Arms 1 and 3 (without and with co-administration of DLM). AUC 0-22h defines area under the concentration-time curve over the period of 22 hours post-dose.
Time Frame: Intensive BDQ PK samples at pre-dose, 5h, 7h, 10h and 22h post-dose at Weeks 2, 8 and 24
Population: Participants who took at least one dose of study treatment, and were taking study drug at the time of the PK visit.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Arm 1: Bedaquiline | Arm 3: Bedaquiline and Delamanid
Number analyzed (Participants) | 28 | 24
ng*h/mL
  Week 2 | 31570.9 (14612.8) | 32399.4 (13625.2)
  Week 8: number analyzed (Participants) | 25 | 21
  Week 8 | 19234.6 (7785.7) | 20176.1 (8175.5)
  Week 24: number analyzed (Participants) | 24 | 18
  Week 24 | 21048.5 (8329.7) | 19522.6 (7545.7)
Statistical Analysis 1: Comparison: Arm 1: Bedaquiline vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 2; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 1.036, 90% CI 2-sided [0.847 to 1.267] — The numerator represents Arm 3 and the denominator represents Arm 1
Statistical Analysis 2: Comparison: Arm 1: Bedaquiline vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 8; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 1.037, 90% CI 2-sided [0.843 to 1.276] — The numerator represents Arm 3 and the denominator represents Arm 1
Statistical Analysis 3: Comparison: Arm 1: Bedaquiline vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 24; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 0.915, 90% CI 2-sided [0.727 to 1.151] — The numerator represents Arm 3 and the denominator represents Arm 1

11. Secondary Outcome: N-monodesmethyl Metabolite of BDQ PK Parameter Cmin Determined Based on BDQ Metabolite Levels From Individual Participants Enrolled in Arms 1 and 3
Description: This evaluates the effect of DLM on the N-monodesmethyl Metabolite of BDQ PK parameter Cmin obtained from participants enrolled in Arms 1 and 3 (without and with co-administration of DLM). Cmin defines minimum concentration observed over the first 22 hours of the BDQ dosing interval.
Time Frame: Intensive BDQ Metabolite PK samples at pre-dose, 5h, 7h, 10h and 22h post-dose at weeks 2, 8 and 24
Population: Participants who took at least one dose of study treatment, and were taking study drug at the time of the PK visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1: Bedaquiline | Arm 3: Bedaquiline and Delamanid
Number analyzed (Participants) | 28 | 26
ng/mL
  Week 2 | 353.3 (137.8) | 361.6 (122.8)
  Week 8: number analyzed (Participants) | 25 | 23
  Week 8 | 200.0 (81.1) | 204.7 (76.3)
  Week 24: number analyzed (Participants) | 24 | 20
  Week 24 | 204.0 (62.8) | 174.0 (82.1)
Statistical Analysis 1: Comparison: Arm 1: Bedaquiline vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 2; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 1.043, 90% CI 2-sided [0.864 to 1.258] — The numerator represents Arm 3 and the denominator represents Arm 1
Statistical Analysis 2: Comparison: Arm 1: Bedaquiline vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 8; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 1.029, 90% CI 2-sided [0.858 to 1.235] — The numerator represents Arm 3 and the denominator represents Arm 1
Statistical Analysis 3: Comparison: Arm 1: Bedaquiline vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 24; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 0.808, 90% CI 2-sided [0.657 to 0.993] — The numerator represents Arm 3 and the denominator represents Arm 1

12. Secondary Outcome: N-monodesmethyl Metabolite of BDQ PK Parameter Cmax Determined Based on BDQ Metabolite Levels From Individual Participants Enrolled in Arms 1 and 3
Description: This evaluates the effect of DLM on the BDQ Metabolite N-monodesmethyl BDQ PK parameter Cmax obtained from participants enrolled in Arms 1 and 3 (without and with co-administration of DLM). Cmax defines maximum concentration observed over the first 22 hours of the BDQ dosing interval.
Time Frame: Intensive BDQ Metabolite PK samples at pre-dose, 5h, 7h, 10h and 22h post-dose at weeks 2, 8 and 24
Population: Participants who took at least one dose of study treatment, and were taking study drug at the time of the PK visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1: Bedaquiline | Arm 3: Bedaquiline and Delamanid
Number analyzed (Participants) | 28 | 26
ng/mL
  Week 2 | 404.8 (143.7) | 429.8 (139.8)
  Week 8: number analyzed (Participants) | 25 | 23
  Week 8 | 248.5 (95.4) | 241.5 (87.2)
  Week 24: number analyzed (Participants) | 24 | 20
  Week 24 | 232.9 (68.6) | 196.8 (92.5)
Statistical Analysis 1: Comparison: Arm 1: Bedaquiline vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 2; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 1.068, 90% CI 2-sided [0.903 to 1.263] — The numerator represents Arm 3 and the denominator represents Arm 1
Statistical Analysis 2: Comparison: Arm 1: Bedaquiline vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 8; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 0.973, 90% CI 2-sided [0.820 to 1.155] — The numerator represents Arm 3 and the denominator represents Arm 1
Statistical Analysis 3: Comparison: Arm 1: Bedaquiline vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 24; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 0.803, 90% CI 2-sided [0.656 to 0.983] — The numerator represents Arm 3 and the denominator represents Arm 1

13. Secondary Outcome: N-monodesmethyl Metabolite of BDQ PK Parameter AUC 0-22h Calculated Based on Intensive PK Samples Obtained From Individual Participants Enrolled in Arms 1 and 3
Description: This evaluates the effect of DLM on the N-monodesmethyl Metabolite of BDQ PK parameter AUC 0-22h obtained from participants enrolled in Arms 1 and 3 (without and with co-administration of DLM). AUC 0-22h defines area under the concentration-time curve over the period of 22 hours post-dose.
Time Frame: Intensive BDQ PK samples at pre-dose, 5h, 7h, 10h and 22h post-dose at Weeks 2, 8 and 24
Population: Participants who took at least one dose of study treatment, and were taking study drug at the time of the PK visit.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Arm 1: Bedaquiline | Arm 3: Bedaquiline and Delamanid
Number analyzed (Participants) | 28 | 26
ng*h/mL
  Week 2 | 8435.5 (3220.1) | 8713.4 (2858.9)
  Week 8: number analyzed (Participants) | 25 | 23
  Week 8 | 5067.5 (2017.6) | 4963.4 (1847.6)
  Week 24: number analyzed (Participants) | 24 | 20
  Week 24 | 4771.4 (1577.9) | 4033.5 (1978.7)
Statistical Analysis 1: Comparison: Arm 1: Bedaquiline vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 2; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 1.049, 90% CI 2-sided [0.881 to 1.248] — The numerator represents Arm 3 and the denominator represents Arm 1
Statistical Analysis 2: Comparison: Arm 1: Bedaquiline vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 8; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 0.979, 90% CI 2-sided [0.823 to 1.165] — The numerator represents Arm 3 and the denominator represents Arm 1
Statistical Analysis 3: Comparison: Arm 1: Bedaquiline vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 24; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 0.808, 90% CI 2-sided [0.638 to 1.025] — The numerator represents Arm 3 and the denominator represents Arm 1

14. Secondary Outcome: DLM PK Parameter Cmin Determined Based on DLM Levels From Individual Participants Enrolled in Arms 2 and 3
Description: This evaluates the effect of BDQ on the DLM PK parameter Cmin obtained from participants enrolled in Arms 2 and 3 (without and with co-administration of BDQ). Cmin defines minimum concentration observed over the first 11 hours of the DLM dosing interval.
Time Frame: Intensive DLM PK samples at pre-dose, 4h, 8h, and 11h post-dose at weeks 2, 8 and 24
Population: Participants who took at least one dose of study treatment, and were taking study drug at the time of the PK visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 2: Delamanid | Arm 3: Bedaquiline and Delamanid
Number analyzed (Participants) | 25 | 26
ng/mL
  Week 2 | 224.8 (59.0) | 206.8 (64.8)
  Week 8: number analyzed (Participants) | 24 | 24
  Week 8 | 198.2 (64.3) | 217.2 (64.6)
  Week 24: number analyzed (Participants) | 20 | 19
  Week 24 | 220.9 (78.9) | 182.2 (78.5)
Statistical Analysis 1: Comparison: Arm 2: Delamanid vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 2; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 0.903, 90% CI 2-sided [0.778 to 1.049] — The numerator represents Arm 3 and the denominator represents Arm 2
Statistical Analysis 2: Comparison: Arm 2: Delamanid vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 8; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 1.114, 90% CI 2-sided [0.944 to 1.315] — The numerator represents Arm 3 and the denominator represents Arm 2
Statistical Analysis 3: Comparison: Arm 2: Delamanid vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 24; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 0.804, 90% CI 2-sided [0.639 to 1.012] — The numerator represents Arm 3 and the denominator represents Arm 2

15. Secondary Outcome: DLM PK Parameter Cmax Determined Based on DLM Levels From Individual Participants Enrolled in Arms 2 and 3
Description: This evaluates the effect of BDQ on the DLM PK parameter Cmax obtained from participants enrolled in Arms 2 and 3 (without and with co-administration of BDQ). Cmax defines maximum concentration observed over the first 11 hours of the DLM dosing interval.
Time Frame: Intensive DLM PK samples at pre-dose, 4h, 8h, and 11h post-dose at weeks 2, 8 and 24
Population: Participants who took at least one dose of study treatment, and were taking study drug at the time of the PK visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 2: Delamanid | Arm 3: Bedaquiline and Delamanid
Number analyzed (Participants) | 25 | 26
ng/mL
  Week 2 | 317.8 (88.7) | 298.3 (84.2)
  Week 8: number analyzed (Participants) | 24 | 24
  Week 8 | 294.1 (100.0) | 320.9 (98.4)
  Week 24: number analyzed (Participants) | 20 | 19
  Week 24 | 290.3 (81.6) | 259.0 (102.8)
Statistical Analysis 1: Comparison: Arm 2: Delamanid vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 2; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 0.937, 90% CI 2-sided [0.810 to 1.084] — The numerator represents Arm 3 and the denominator represents Arm 2
Statistical Analysis 2: Comparison: Arm 2: Delamanid vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 8; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 1.107, 90% CI 2-sided [0.929 to 1.318] — The numerator represents Arm 3 and the denominator represents Arm 2
Statistical Analysis 3: Comparison: Arm 2: Delamanid vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 24; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 0.856, 90% CI 2-sided [0.703 to 1.043] — The numerator represents Arm 3 and the denominator represents Arm 2

16. Secondary Outcome: DLM PK Area Under the Concentration Time Curve (AUC 0-11h) Determined Based on Intensive PK Samples Obtained From Individual Participants Enrolled in Arms 2 and 3
Description: This evaluates the effect of BDQ on the DLM PK parameter AUC 0-11h obtained from participants enrolled in Arms 2 and 3 (without and with co-administration of BDQ). AUC 0-11h defines area under the concentration-time curve over the first 11 hours of the DLM dosing interval.
Time Frame: Intensive DLM PK samples at pre-dose, 4h, 8h, and 11h post-dose at weeks 2, 8 and 24
Population: Participants who took at least one dose of study treatment, and were taking study drug at the time of the PK visit.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Arm 2: Delamanid | Arm 3: Bedaquiline and Delamanid
Number analyzed (Participants) | 25 | 26
ng*h/mL
  Week 2 | 2789.6 (761.9) | 2654.9 (724.3)
  Week 8: number analyzed (Participants) | 24 | 24
  Week 8 | 2547.6 (838.4) | 2823.2 (792.7)
  Week 24: number analyzed (Participants) | 20 | 19
  Week 24 | 2473.0 (778.2) | 2324.9 (987.3)
Statistical Analysis 1: Comparison: Arm 2: Delamanid vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 2; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 0.951, 90% CI 2-sided [0.825 to 1.096] — The numerator represents Arm 3 and the denominator represents Arm 2
Statistical Analysis 2: Comparison: Arm 2: Delamanid vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 8; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 1.136, 90% CI 2-sided [0.948 to 1.362] — The numerator represents Arm 3 and the denominator represents Arm 2
Statistical Analysis 3: Comparison: Arm 2: Delamanid vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 24; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 0.898, 90% CI 2-sided [0.727 to 1.109] — The numerator represents Arm 3 and the denominator represents Arm 2

17. Secondary Outcome: DLM Metabolite DM6705 PK Parameter Cmin Determined Based on DLM Metabolite Levels From Individual Participants Enrolled in Arms 2 and 3
Description: This evaluates the effect of BDQ on the DLM Metabolite DM6705 PK parameter Cmin obtained from participants enrolled in Arms 2 and 3 (without and with co-administration of BDQ). Cmin defines minimum concentration observed over the first 11 hours of the DLM dosing interval.
Time Frame: Intensive DLM PK samples at pre-dose, 4h, 8h, and 11h post-dose at weeks 2, 8 and 24
Population: Participants who took at least one dose of study treatment, and were taking study drug at the time of the PK visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 2: Delamanid | Arm 3: Bedaquiline and Delamanid
Number analyzed (Participants) | 25 | 26
ng/mL
  Week 2 | 61.9 (19.3) | 58.5 (17.0)
  Week 8: number analyzed (Participants) | 24 | 24
  Week 8 | 90.6 (38.2) | 94.4 (37.8)
  Week 24: number analyzed (Participants) | 20 | 19
  Week 24 | 75.7 (41.6) | 71.0 (46.6)
Statistical Analysis 1: Comparison: Arm 2: Delamanid vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 2; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 0.939, 90% CI 2-sided [0.806 to 1.094] — The numerator represents Arm 3 and the denominator represents Arm 2
Statistical Analysis 2: Comparison: Arm 2: Delamanid vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 8; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 1.081, 90% CI 2-sided [0.864 to 1.352] — The numerator represents Arm 3 and the denominator represents Arm 2
Statistical Analysis 3: Comparison: Arm 2: Delamanid vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 24; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 0.865, 90% CI 2-sided [0.597 to 1.253] — The numerator represents Arm 3 and the denominator represents Arm 2

18. Secondary Outcome: DLM Metabolite DM6705 PK Parameter Cmax Determined Based on DLM Metabolite Levels From Individual Participants Enrolled in Arms 2 and 3
Description: This evaluates the effect of BDQ on the DLM Metabolite DM6705 PK parameter Cmax obtained from participants enrolled in Arms 2 and 3 (without and with co-administration of BDQ). Cmax defines maximum concentration observed over the first 11 hours of the DLM dosing interval.
Time Frame: Intensive DLM PK samples at pre-dose, 4h, 8h, and 11h post-dose at weeks 2, 8 and 24
Population: Participants who took at least one dose of study treatment, and were taking study drug at the time of the PK visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 2: Delamanid | Arm 3: Bedaquiline and Delamanid
Number analyzed (Participants) | 25 | 26
ng/mL
  Week 2 | 66.6 (18.1) | 64.3 (19.8)
  Week 8: number analyzed (Participants) | 24 | 24
  Week 8 | 99.7 (41.0) | 105.4 (46.2)
  Week 24: number analyzed (Participants) | 20 | 19
  Week 24 | 82.1 (46.1) | 75.6 (47.9)
Statistical Analysis 1: Comparison: Arm 2: Delamanid vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 2; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 0.950, 90% CI 2-sided [0.825 to 1.095] — The numerator represents Arm 3 and the denominator represents Arm 2
Statistical Analysis 2: Comparison: Arm 2: Delamanid vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 8; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 1.080, 90% CI 2-sided [0.862 to 1.354] — The numerator represents Arm 3 and the denominator represents Arm 2
Statistical Analysis 3: Comparison: Arm 2: Delamanid vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 24; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 0.865, 90% CI 2-sided [0.605 to 1.239] — The numerator represents Arm 3 and the denominator represents Arm 2

19. Secondary Outcome: DLM Metabolite DM6705 PK AUC 0-11h Determined Based on Intensive PK Samples Obtained From Individual Participants Enrolled in Arms 2 and 3
Description: This evaluates the effect of BDQ on the DLM Metabolite DM6705 PK parameter AUC 0-11h obtained from participants enrolled in Arms 2 and 3 (without and with co-administration of BDQ). AUC 0-11h defines area under the concentration-time curve over the first 11 hours of the DLM dosing interval.
Time Frame: Intensive DLM PK samples at pre-dose, 4h, 8h, and 11h post-dose at weeks 2, 8 and 24
Population: Participants who took at least one dose of study treatment, and were taking study drug at the time of the PK visit.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Arm 2: Delamanid | Arm 3: Bedaquiline and Delamanid
Number analyzed (Participants) | 25 | 26
ng*h/mL
  Week 2 | 628.0 (188.1) | 621.2 (178.3)
  Week 8: number analyzed (Participants) | 24 | 24
  Week 8 | 953.9 (395.2) | 990.9 (378.1)
  Week 24: number analyzed (Participants) | 20 | 19
  Week 24 | 749.9 (420.4) | 742.5 (479.5)
Statistical Analysis 1: Comparison: Arm 2: Delamanid vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 2; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 0.984, 90% CI 2-sided [0.851 to 1.138] — The numerator represents Arm 3 and the denominator represents Arm 2
Statistical Analysis 2: Comparison: Arm 2: Delamanid vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 8; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 1.086, 90% CI 2-sided [0.866 to 1.361] — The numerator represents Arm 3 and the denominator represents Arm 2
Statistical Analysis 3: Comparison: Arm 2: Delamanid vs Arm 3: Bedaquiline and Delamanid; Statistical analysis for Week 24; Test type: Equivalence — GMRs were compared to no effect boundaries of 0.67 to 1.50; Geometric Mean Ratio = 0.927, 90% CI 2-sided [0.650 to 1.322] — The numerator represents Arm 3 and the denominator represents Arm 2

20. Secondary Outcome: Percentage of Participants With an Occurrence of Grade 3 or Higher Adverse Event
Description: Participants with an occurrence of an adverse event (laboratory value, sign/symptom, diagnosis) of grade 3 or 4. Severity grading based on DAIDS AE Grading Table Version 2.0. Participants were counted once at the highest grade (grade 3 or grade 4).
Time Frame: From initiation of study TB treatment (week 0) to week 24
Population: Participants who took at least one dose of study TB treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: Bedaquiline | Arm 2: Delamanid | Arm 3: Bedaquiline and Delamanid
Number analyzed (Participants) | 28 | 27 | 27
Percentage of participants
  Grade 3 adverse event | 36 [19 to 56] | 11 [2 to 29] | 19 [6 to 38]
  Grade 4 adverse event | 4 [0 to 18] | 11 [2 to 29] | 19 [6 to 38]

21. Secondary Outcome: Percentage of Participants Who Discontinued Study TB Drug(s) For Any Reason
Description: Percentage of participants who discontinued study TB drug(s) for any reason
Time Frame: From initiation of study TB treatment (week 0) to week 24
Population: Participants who took at least one dose of study TB treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: Bedaquiline | Arm 2: Delamanid | Arm 3: Bedaquiline and Delamanid
Number analyzed (Participants) | 28 | 27 | 27
Percentage of participants | 11 [2 to 28] | 19 [6 to 38] | 22 [9 to 42]

22. Secondary Outcome: Percentage of Participants Who Died
Description: Among participants who took at least one dose of study TB treatment, percentage of participants who died on or before week 24. Note that the all-cause mortality includes deaths that occurred at any time during treatment or follow-up through week 128.
Time Frame: From initiation of study TB treatment (week 0) to week 24
Population: Participants who took at least one dose of study TB treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: Bedaquiline | Arm 2: Delamanid | Arm 3: Bedaquiline and Delamanid
Number analyzed (Participants) | 28 | 27 | 27
Percentage of participants | 0 [0 to 12] | 0 [0 to 13] | 0 [0 to 13]

ADVERSE EVENTS:
Time Frame: From start of study treatment to study completion at Week 128 or premature study discontinuation.
Description: For participants who took at least one dose of study TB treatment. All diagnoses (per ACTG criteria for clinical events and other diseases); signs/symptoms (S/S) of grade 3 or higher or any S/S that led to a change in BDQ, DLM and/or DTG regardless of grade; hematologies, LFTs and chemistries of grade 3 and higher, or any laboratory finding that led to a change in BDQ, DLM and/or DTG regardless of grade.The DAIDS AE Grading Table Version 2.0, and the DAIDS EAE Manual Version 2.0 were used.
Arm/Group | Arm 1: Bedaquiline | Arm 2: Delamanid | Arm 3: Bedaquiline and Delamanid
All-Cause Mortality (participants affected / at risk) | 0/28 | 1/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 2/28 | 3/27 | 8/27
Other Adverse Events (participants affected / at risk) | 21/28 | 16/27 | 21/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Bedaquiline (N=28) | Arm 2: Delamanid (N=27) | Arm 3: Bedaquiline and Delamanid (N=27)
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Stab wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 4
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Focal dyscognitive seizures (Nervous system disorders) | 0 | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Bedaquiline (N=28) | Arm 2: Delamanid (N=27) | Arm 3: Bedaquiline and Delamanid (N=27)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 1
Deafness (Ear and labyrinth disorders) | 3 | 2 | 6
Deafness neurosensory (Ear and labyrinth disorders) | 8 | 4 | 4
Tinnitus (Ear and labyrinth disorders) | 2 | 0 | 2
Conjunctivitis allergic (Eye disorders) | 0 | 2 | 1
Optic neuropathy (Eye disorders) | 0 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 3 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 3
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0
Injection site reaction (General disorders) | 0 | 2 | 0
Acute sinusitis (Infections and infestations) | 1 | 3 | 1
Oral candidiasis (Infections and infestations) | 0 | 6 | 1
Oral herpes (Infections and infestations) | 1 | 2 | 0
Pharyngitis (Infections and infestations) | 3 | 5 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 1
Blood albumin decreased (Investigations) | 1 | 2 | 0
Blood glucose decreased (Investigations) | 0 | 1 | 2
Blood uric acid increased (Investigations) | 3 | 1 | 0
Haemoglobin decreased (Investigations) | 3 | 0 | 1
Weight decreased (Investigations) | 3 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1
Dizziness (Nervous system disorders) | 3 | 0 | 2
Headache (Nervous system disorders) | 3 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 6 | 2 | 3
Paraesthesia (Nervous system disorders) | 4 | 1 | 2
Seizure (Nervous system disorders) | 0 | 0 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 8 | 6 | 8
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Hypertension (Vascular disorders) | 2 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/48/NCT02583048/Prot_001.pdf
  • Statistical Analysis Plan (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/48/NCT02583048/SAP_000.pdf